CLINICAL TRIAL: NCT01696383
Title: Assessing the Efficacy of DuoTrav® (Travoprost 0.004%/Timolol 0.5% Fixed Combination), as a Replacement Therapy in Glaucoma Patients in Russia, Previously on Prior Prostaglandin Analogue or Beta-blocker Monotherapy
Brief Title: Assessing the Efficacy of DuoTrav as a Replacement Therapy in Glaucoma Patients in Russia
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Management decision
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RDG-11-257
Record Dates: First submitted 2012-09-27; First posted 2012-10-01 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: Intraocular Pressure (IOP); Glaucoma; Ocular hypertension; DuoTrav; Prostaglandin analogue; Beta-blocker
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Travoprost; Timolol; Duotrav

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DuoTrav (Experimental): One drop self-administered topically to the study eye(s) once daily every evening at 8:00 pm for 12 weeks
  Interventions: Drug: Travoprost 0.004%/Timolol 0.5% Fixed Combination (DuoTrav)

INTERVENTIONS:
Drug: Travoprost 0.004%/Timolol 0.5% Fixed Combination (DuoTrav) — One drop self-administered topically to the study eye(s) once daily every evening at 8:00 pm for 12 weeks
  Other Names: DuoTrav®

SUMMARY:
The purpose of this study is to evaluate the efficacy of changing to DuoTrav® (Travoprost 0.004%/Timolol 0.5%) from prior prostaglandin analogue or beta-blocker monotherapy in Russian glaucoma patients with open-angle glaucoma or ocular hypertension whose intraocular pressure (IOP) is uncontrolled while on their current treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ocular hypertension, primary open-angle glaucoma and pseudoexfoliative or pigment dispersion glaucoma.
* Be on a stable IOP-lowering regimen of prostaglandin analogue or beta-blocker (monotherapy) within 4 weeks prior to the Screening Visit.
* Have IOP considered to be safe (in the opinion of the investigator), in both eyes, in such a way that should assure clinical stability of vision and the optic nerve throughout the study period.
* Have an IOP of between 19 to 35 mmHg (at any time of the day) in at least one eye (which would be designated as the study eye). In any eye not designated as a study eye, the IOP should be able to be controlled on no pharmacologic therapy or on the study medicine alone.
* Willing to discontinue the use of all other ocular hypotensive medication(s) prior to receiving the study medication for the entire course of the study.
* Able to follow instructions and willing and able to attend all study visits.
* Have best corrected visual acuity of 6/60 (20/200 Snellen, 1.0 LogMAR) or better in each eye.
* Read, sign, and date an Ethics Committee reviewed and approved informed consent form.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Known medical history of allergy, hypersensitivity or poor tolerance to any component of DuoTrav® that is deemed clinically significant in the opinion of the Principal Investigator.
* Any abnormality preventing reliable applanation tonometry in either eye.
* Corneal dystrophies in either eye.
* Any opacity or subject uncooperativeness that restricts adequate examination of the anterior chamber of either eye.
* Concurrent infectious/noninfectious conjunctivitis, keratitis or uveitis in either eye. Blepharitis or non-clinically significant conjunctival injection is allowed.
* History of ocular herpes simplex infection.
* Intraocular conventional surgery or laser surgery in either eye that is less than three months prior to the Screening Visit.
* Risk of visual field or visual acuity worsening as a consequence of participation in the study, in the investigator's best judgment.
* Progressive retinal or optic nerve disease from any cause apart from glaucoma.
* Use of systemic medications known to affect IOP (e.g., oral beta-adrenergic blockers, alpha-agonists and blockers, angiotensin converting enzyme inhibitors and calcium channel blockers), which have not been on a stable course for 7 days prior to Screening Visit or an anticipated change in the dosage during the course of the study.
* Bronchial asthma, a history of bronchial asthma, or severe chronic obstructive pulmonary disease that would preclude the safe administration of a topical beta-blocker.
* History of severe allergic rhinitis.
* Unwillingness to risk the possibility of darkened iris or eyelash changes.
* Women of childbearing potential not using reliable means of birth control for at least one month prior to the Screening/Baseline Visit.
* Women who are pregnant or lactating.
* Participation in any other investigational study within 30 days prior to the Screening Visit.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline (Day 0) in intraocular pressure (IOP) at final visit (Week 12) | Baseline (Day 0), Week 12
  As measured by Goldmann applanation tonometry. If only one eye qualifies for inclusion and treatment, this eye will be selected for analysis. If both eyes qualify and are treated, the worse evaluable eye will be selected for analysis. The worse eye will be the eye with the higher IOP at the screening/baseline visit. If both eyes are equal, the right eye will be selected for analysis.

SECONDARY OUTCOMES:
Percentage of subjects who reach target IOP (≤18 mmHg) | Week 12
  As measured by Goldmann applanation tonometry.

CONTACTS AND LOCATIONS:
Overall Officials: Abayomi Ogundele, PharmD, Study Director — Alcon Research